CLINICAL TRIAL: NCT07328035
Title: Remission in Adults With Severe Asthma in Thailand
Status: Not yet recruiting | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Associate Professor, Thammasat University
Other Study IDs: MTU-EC-IM-0-283/68
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Severe Asthma; Asthma Control Level
Keywords: asthma; remission; Thailand; severe; FeNO; blood eosinophil count
MeSH Terms: conditions — Asthma; Lymphoma, Follicular | interventions — Surveys and Questionnaires; Spirometry; Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe asthma: Asthma that requires treatment with high-dose inhaled corticosteroids plus a second controller, or requires systemic corticosteroids for ≥50% of the previous year to prevent it from becoming uncontrolled, or remains uncontrolled despite this therapy.
  Interventions: Other: Global Initiative for Asthma (GINA) and Asthma Control Test (ACT) questionnaires; Diagnostic Test: Spirometry; Diagnostic Test: Fractional exhaled nitric oxide (FeNO) test; Diagnostic Test: Blood eosinophil count (BEC)

INTERVENTIONS:
Other: Global Initiative for Asthma (GINA) and Asthma Control Test (ACT) questionnaires — GINA and ACT are questionnaires used to assess the level of asthma control.
Diagnostic Test: Spirometry — Spirometry is a tool used to assess pulmonary function.
Diagnostic Test: Fractional exhaled nitric oxide (FeNO) test — FeNO is a tool used to assess eosinophilic airway inflammation and asthma remission.
Diagnostic Test: Blood eosinophil count (BEC) — BEC is a tool used to assess eosinophilic inflammation and asthma remission.

SUMMARY:
The goal of this observational study is to determine the prevalence of remission among adults with severe asthma, as well as the factors associated with remission in Thailand.

The main question the study aims to answer is:

What is the prevalence of remission among adults with severe asthma in Thailand? Participants will complete questionnaires on asthma symptoms and undergo pulmonary function testing and a blood test once.

DETAILED DESCRIPTION:
This study is a cross-sectional study. Thai patients aged 18 years or older with severe asthma are included in the study. Participants will complete two questionnaires about asthma control: the Global Initiative for Asthma (GINA) and the Asthma Control Test (ACT), and will perform spirometry, a fractional exhaled nitric oxide (FeNO) test, and blood eosinophil counts (BEC).

ELIGIBILITY:
Inclusion Criteria:

* severe asthma
* age 18 years or older

Exclusion Criteria:

* inability to perform spirometry or fractional exhaled nitric oxide (FeNO) test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thai patients aged 18 years or older with severe asthma are included in the study
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence rate of severe asthma remission | The beginning of the study
  Prevalence rate of remission in adults with severe asthma

SECONDARY OUTCOMES:
Association of clinical characteristics with severe asthma remission | The beginning of the study
  The association between severe asthma remission and the following variables will be evaluated:
  1. Asthma symptom control; Asthma Control Test (ACT) score (range 5-25)
  2. Exacerbation history; Number of asthma exacerbations requiring systemic corticosteroids in the previous 12 months
  3. Oral corticosteroid use; Daily oral corticosteroid use (yes/no) and cumulative dose (mg/year)
  4. Asthma duration; Years since asthma diagnosis
Association of lung function with severe asthma remission | The beginning of the study
  The association between severe asthma remission (binary outcome: remission vs. non-remission) and pulmonary function assessed using spirometry (FEV1 % predicted and FEV1/FVC ratio).
Association of inflammatory biomarkers with severe asthma remission | The beginning of the study
  The association between severe asthma remission (binary outcome: remission vs. non-remission) and inflammatory biomarkers assessed using blood eosinophil count (cells/µL) and fractional exhaled nitric oxide (FeNO) (parts per billion, ppb).

CONTACTS AND LOCATIONS:
Overall Officials: Narongkorn Saiphoklang, Principal Investigator — Thammasat University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: Yes
IPD and documents
Supporting Information: Study Protocol, SAP
Time Frame: IPD and documents will be available for sharing immediately after publication for a period of 2 years.

REFERENCES:
- [Result] McDowell PJ, McDowell R, Busby J, Eastwood MC, Patel PH, Jackson DJ, Mansur A, Patel M, Burhan H, Doe S, Chaudhuri R, Gore R, Dodd JW, Subramanian D, Brown T, Heaney LG; UK Severe Asthma Registry. Clinical remission in severe asthma with biologic therapy: an analysis from the UK Severe Asthma Registry. Eur Respir J. 2023 Dec 14;62(6):2300819. doi: 10.1183/13993003.00819-2023. Print 2023 Dec. PMID 37857423
- [Result] Tupper OD, Hakansson KEJ, Ulrik CS. Remission and Changes in Severity Over 30 Years in an Adult Asthma Cohort. J Allergy Clin Immunol Pract. 2021 Apr;9(4):1595-1603.e5. doi: 10.1016/j.jaip.2020.11.013. Epub 2020 Nov 19. PMID 33220516
- [Result] Chipps BE, Lugogo N, Carr W, Zhou W, Patel A, Carstens DD, Trudo F, Ambrose CS. On-treatment clinical remission of severe asthma with real-world longer-term biologic use. J Allergy Clin Immunol Glob. 2024 Oct 30;4(1):100365. doi: 10.1016/j.jacig.2024.100365. eCollection 2025 Feb. PMID 39659738
- [Result] Perez-de-Llano L, Scelo G, Tran TN, Le TT, Fageras M, Cosio BG, Peters M, Pfeffer PE, Al-Ahmad M, Al-Lehebi RO, Altraja A, Bergeron C, Bjermer LH, Bjerrum AS, Bulathsinhala L, Busby J, Cano Rosales DJ, Canonica GW, Carter VA, Charriot J, Christoff GC, Denton EJ, Dorscheid DR, Fernandez Sanchez MJ, Fonseca JA, Gibson PG, Goh CYY, Heaney LG, Heffler E, Hew M, Iwanaga T, Katial R, Koh MS, Kuna P, Larenas-Linnemann DES, Lehtimaki L, Mahboub B, Martin N, Matsumoto H, Menzies-Gow AN, Papadopoulos NG, Popov TA, Porsbjerg CM, Patel P, Rhee CK, Sadatsafavi M, Taille C, Torres-Duque CA, Tsai MJ, Ulrik CS, Upham JW, von Bulow A, Wang E, Wechsler ME, Price DB. Exploring Definitions and Predictors of Severe Asthma Clinical Remission after Biologic Treatment in Adults. Am J Respir Crit Care Med. 2024 Oct 1;210(7):869-880. doi: 10.1164/rccm.202311-2192OC. PMID 38701495
- [Result] Hansen S, Baastrup Sondergaard M, von Bulow A, Bjerrum AS, Schmid J, Rasmussen LM, Johnsen CR, Ingebrigtsen T, Hakansson KEJ, Johansson SL, Bisgaard M, Assing KD, Hilberg O, Ulrik C, Porsbjerg C. Clinical Response and Remission in Patients With Severe Asthma Treated With Biologic Therapies. Chest. 2024 Feb;165(2):253-266. doi: 10.1016/j.chest.2023.10.046. Epub 2023 Nov 3. PMID 37925144
- [Result] Holm M, Omenaas E, Gislason T, Svanes C, Jogi R, Norrman E, Janson C, Toren K; RHINE Study Group. Remission of asthma: a prospective longitudinal study from northern Europe (RHINE study). Eur Respir J. 2007 Jul;30(1):62-5. doi: 10.1183/09031936.00121705. Epub 2007 Mar 14. PMID 17360725
- [Result] Almqvist L, Ronmark E, Stridsman C, Backman H, Lindberg A, Lundback B, Hedman L. Remission of adult-onset asthma is rare: a 15-year follow-up study. ERJ Open Res. 2020 Nov 23;6(4):00620-2020. doi: 10.1183/23120541.00620-2020. eCollection 2020 Oct. PMID 33263024